CLINICAL TRIAL: NCT00899704
Title: Molecular Mechanisms of OSCC Tumor Invasion
Brief Title: Biomarkers in Tissue Samples From Patients Who Have Undergone Neck Dissection for Oral Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study was never published
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z3081; ACOSOG-Z3081; CDR0000589332 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Tongue Neoplasms | interventions — Microarray Analysis; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patient tissue samples are screened using polymerase chain reaction (PCR) for human papilloma virus-specific primers. Samples are analyzed to identify a nodal-metastasis signature for oral squamous cell carcinoma. Samples also undergo microarray analysis to quantify expression levels for targeted genes. Initial data analysis is performed using Affymetrix® Microarray Suite 5.0 to quantify expression levels for targeted genes.
  Interventions: Genetic: microarray analysis; Genetic: allele-specific oligonucleotide real-time quantitative polymerase chain reaction; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Genetic: microarray analysis
  Other Names: gene expression profiling
Genetic: allele-specific oligonucleotide real-time quantitative polymerase chain reaction
  Other Names: ASO RQ-PCR
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tissue samples in predicting oral cancer in patients who have undergone neck dissection for oral cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test preliminary data from node-positive oral squamous cell carcinoma (OSCC) signatures for their ability to predict lymph-positive primaries using a cohort of OSCC tumors.
* To perform lymph node prediction using sentinel lymph node-biopsied primaries.
* To validate the preliminary data node-positive OSCC signature and test its ability to predict nodal status.

OUTLINE: Patient tissue samples are screened using polymerase chain reaction (PCR) for human papilloma virus-specific primers. Samples are analyzed to identify a nodal-metastasis signature for oral squamous cell carcinoma. Samples also undergo microarray analysis to quantify expression levels for targeted genes. Initial data analysis is performed using Affymetrix® Microarray Suite 5.0 to quantify expression levels for targeted genes.

ELIGIBILITY:
* Have a primary tumor specimen banked by the American College of Surgeons Oncology Group (ACOSOG) as part of clinical trial ACOSOG-Z0360

  * All tumor specimens are squamous cell carcinomas of the tongue, floor of the mouth, or gingiva
* All patients have undergone neck dissections * Pathologically confirmed nodal stage (negative or positive)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient tissue samples are screened using polymerase chain reaction (PCR) for human papilloma virus-specific primers. Samples are analyzed to identify a nodal-metastasis signature for oral squamous cell carcinoma. Samples also undergo microarray analysis to quantify expression levels for targeted genes. Initial data analysis is performed using Affymetrix® Microarray Suite 5.0 to quantify expression levels for targeted genes. are
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Barry Ziober, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States